CLINICAL TRIAL: NCT01335308
Title: Brief Motivational Interviewing to Reduce Child Body Mass Index
Acronym: BMi2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Academy of Pediatrics (Other); Academy of Nutrition and Dietetics (Other); University of Iowa (Other)
Responsible Party: Principal Investigator, Ken Resnicow, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HL085400; 5R01HL085400 (NIH)
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Childhood Obesity
Keywords: Pediatric Obesity; Motivational Interviewing; Overweight; Behavior Change
MeSH Terms: conditions — Pediatric Obesity; Overweight | interventions — Standard of Care; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Care with Education Materials (Active Comparator): Measure height and weight only. usual care
  Interventions: Behavioral: Standard Care
- Moderate Dose Motivational Interviewing (Experimental): MI delivered by PCP, 4 sessions
  Interventions: Behavioral: Moderate Dose Motivational Interviewing
- Higher Dose Motivational Interviewing (Experimental): MI delivered by PCP, 4 sessions plus MI delivered by RD, 6 sessions
  Interventions: Behavioral: Higher Dose Motivational Interviewing

INTERVENTIONS:
Behavioral: Standard Care — Practitioners will receive 2 hour obesity lecture and ½ day protocol training. Families recruited are given parent education materials. Outcomes will be collected at 1 year and 2 years after enrollment
  Arms: Standard Care with Education Materials
Behavioral: Moderate Dose Motivational Interviewing — Practitioners receive 2 days of Motivational Interviewing and Behavioral Therapy Training and ½ day protocol training. Families recruited receive 4 x MI visits with the pediatric practitioner. Outcomes will be collected at 1 year and 2 years after enrollment
  Arms: Moderate Dose Motivational Interviewing
Behavioral: Higher Dose Motivational Interviewing — Practitioners receive 2 days of Motivational Interviewing and Behavioral Therapy Training and ½ day protocol training. Families recruited receive 4 x MI visits with the pediatric practitioner and 6 x visits (in phone or in person) with a Registered Dietitian, also trained in Motivational Interviewing. Outcomes will be collected at 1 year and 2 years after enrollment
  Arms: Higher Dose Motivational Interviewing

SUMMARY:
BMi 2 is a study that tests a behavioral counseling approach to reduce obesity in children. Practitioners (Pediatricians, Nurse Practitioners) were randomly assigned to one of three groups. The first group continued with standard care; in group 2, each practitioner delivered four study Motivational Interviewing visits with the parent/caregiver, and in group 3 in addition to the practitioner, a registered dietitian delivered 6 Motivational Interviewing visits. The primary outcome will be the child's percentile BMI change between the baseline and 2-year follow-up. Secondary outcomes will include behavior change around fruits and vegetables, sweetened beverages and exercise. Our hypothesis is that there will be a larger decrease in BMI percentile for children in group 3 than in group 2, and that children in group 2 will have a decrease in BMI percentile when compared to group one.

DETAILED DESCRIPTION:
The study is a cluster-randomized intervention trial with clinical practices serving as the unit of randomization and analysis. The investigators are testing two increasingly intensive interventions compared to a minimal intensity/Usual Care Group. Group 1 (Usual Care) includes determination of BMI percentile at baseline, 1-year, and 2-year follow-up. Usual Care (UC) practitioners provide parents with educational materials and routine care. UC pediatricians and their study staff received a ½ day study orientation session which included a brief CME-type workshop addressing obesity treatment.. Group 2 (Pediatric Practitioner only) includes the same assessment points as UC. In addition, Group 2 Pediatric Practitioners (PPs) received 2 days of in-person training in Motivational Interviewing (MI) and Behavior Therapy (BT) as well as an interactive DVD MI booster training system focusing on pediatric obesity. PPs in Group 2 are asked to schedule 3 proactive counseling sessions with a parent of the index child in Year 1 and one additional "booster" visit in year 2. To guide their counseling they are provided with a food and activity screening tool. In addition, Group 2 practices are provided with educational materials written in a style consistent with Motivational Interviewing and Self Determination Theory. Unlike in Group 1, where all of the educational materials are provided proactively to each parent, in Groups 2 and 3, materials are distributed on a more selective tailored basis depending on parent needs. Group 3 (PP+RD) includes the same intervention components as Group 2, but adds MI-based counseling from a trained and registered dietitian (RD) who is linked to that practice. RDs deliver 6 MI-based counseling sessions over 2 years. The intervention is front loaded with 4 sessions in Year 1 and the remaining 2 in Year 2. The RD sessions are delivered both in-person (required for visit 1) and optionally by telephone or in-person, subsequently. Similar to MDs, RDs received 2.0 days of in-person MI and BT training, and the interactive DVD MI booster training system.

ELIGIBILITY:
Inclusion Criteria:

* 85th - 97th percentile BMI
* parent/care giver ability to converse in English
* working telephone

Exclusion Criteria:

* child under current subspecialty care for overweight/obesity
* child currently taking weight-altering medication (at enrollment)

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 645 (Actual)
Dates: Start 2009-10; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Resnicow, PhD, Principal Investigator — University of Michigan; Richard Wasserman, MD, MPH, Principal Investigator — University of Vermont, American Academy of Pediatrics; Erica Slora, PhD, Principal Investigator — American Academy of Pediatrics; Linda G Snetselaar, PhD, Principal Investigator — University of Iowa; Esther Myers, PhD, Principal Investigator — Academy of Nutrition and Dietetics; Fiona McMaster, MA, MPH, Study Director — University of Michigan; Alison Bocian, MSc, Study Director — American Academy of Pediatrics; Donna Harris, MA, Study Director — American Academy of Pediatrics
Locations (1):
- Pediatric Research in Office Settings, Elk Grove Village, Illinois, United States

REFERENCES:
- [Derived] Woolford SJ, Resnicow K, Davis MM, Nichols LP, Wasserman RC, Harris D, Gebremariam A, Shone L, Fiks AG, Chang T. Cost-effectiveness of a motivational interviewing obesity intervention versus usual care in pediatric primary care offices. Obesity (Silver Spring). 2022 Nov;30(11):2265-2274. doi: 10.1002/oby.23560. PMID 36321279
- [Derived] Resnicow K, Harris D, Wasserman R, Schwartz RP, Perez-Rosas V, Mihalcea R, Snetselaar L. Advances in Motivational Interviewing for Pediatric Obesity: Results of the Brief Motivational Interviewing to Reduce Body Mass Index Trial and Future Directions. Pediatr Clin North Am. 2016 Jun;63(3):539-62. doi: 10.1016/j.pcl.2016.02.008. PMID 27261549
- [Derived] Resnicow K, McMaster F, Bocian A, Harris D, Zhou Y, Snetselaar L, Schwartz R, Myers E, Gotlieb J, Foster J, Hollinger D, Smith K, Woolford S, Mueller D, Wasserman RC. Motivational interviewing and dietary counseling for obesity in primary care: an RCT. Pediatrics. 2015 Apr;135(4):649-57. doi: 10.1542/peds.2014-1880. PMID 25825539
- [Derived] Resnicow K, McMaster F, Woolford S, Slora E, Bocian A, Harris D, Drehmer J, Wasserman R, Schwartz R, Myers E, Foster J, Snetselaar L, Hollinger D, Smith K. Study design and baseline description of the BMI2 trial: reducing paediatric obesity in primary care practices. Pediatr Obes. 2012 Feb;7(1):3-15. doi: 10.1111/j.2047-6310.2011.00001.x. Epub 2011 Dec 13. PMID 22434735

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care With Education Materials | Moderate Dose Motivational Interviewing | Higher Dose Motivational Interviewing
Started | 198 | 212 | 235
Completed | 158 | 145 | 154
Not Completed | 40 | 67 | 81

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care With Education Materials | Moderate Dose Motivational Interviewing | Higher Dose Motivational Interviewing | Total
Number analyzed (Participants) | 198 | 212 | 235 | 645
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 198 | 212 | 235 | 645
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 4.7 (1.7) | 5.1 (1.9) | 5.3 (1.8) | 5.1 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 121 | 141 | 367
  Male | 93 | 91 | 94 | 278
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 64 | 49 | 139
  Not Hispanic or Latino | 152 | 139 | 180 | 471
  Unknown or Not Reported | 20 | 9 | 6 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 14 | 3 | 21 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 23 | 14 | 42
  White | 160 | 178 | 188 | 526
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 19 | 8 | 12 | 39
Region of Enrollment [Number; unit: participants]
  United States | 198 | 212 | 235 | 645

OUTCOME MEASURES:

1. Primary Outcome: Child BMI Percentile
Time Frame: 2 years after recruitment
Measure: Mean (Standard Error); unit: BMI Percentile
Arm/Group | Standard Care With Education Materials | Moderate Dose Motivational Interviewing | Higher Dose Motivational Interviewing
Number analyzed (Participants) | 158 | 145 | 154
BMI Percentile | 90.31 (.94) | 88.1 (.94) | 87.1 (.92)

2. Secondary Outcome: Fruit/Vegetable Consumption
Time Frame: 2 years after enrollment
Measure: Mean (Standard Error); unit: Post test adjuste, servings per day
Arm/Group | Standard Care With Education Materials | Moderate Dose Motivational Interviewing | Higher Dose Motivational Interviewing
Number analyzed (Participants) | 158 | 145 | 154
Post test adjuste, servings per day | 3.8 (.12) | 4.1 (.14) | 4.3 (.13)

3. Secondary Outcome: Sweetened Beverage Consumption
Time Frame: 2 years after enrollment
Measure: Mean (Standard Error); unit: Adjusted posted test servings per day
Arm/Group | Standard Care With Education Materials | Moderate Dose Motivational Interviewing | Higher Dose Motivational Interviewing
Number analyzed (Participants) | 158 | 145 | 154
Adjusted posted test servings per day | 1.3 (.11) | 1.3 (.11) | 1.0 (.12)

4. Secondary Outcome: Change in Physical Activity
Time Frame: 2 years after enrollment
Measure: Mean (Standard Error); unit: Adjusted posttest hours per day
Arm/Group | Standard Care With Education Materials | Moderate Dose Motivational Interviewing | Higher Dose Motivational Interviewing
Number analyzed (Participants) | 158 | 145 | 154
Adjusted posttest hours per day | 2.1 (.05) | 1.9 (.06) | 2.1 (.06)

ADVERSE EVENTS:
Arm/Group | Standard Care With Education Materials | Moderate Dose Motivational Interviewing | Higher Dose Motivational Interviewing
Serious Adverse Events (participants affected / at risk) | 0/198 | 0/212 | 0/235
Other Adverse Events (participants affected / at risk) | 0/198 | 0/212 | 0/235

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No